CLINICAL TRIAL: NCT02479399
Title: Specified Drug Use resulTs survEy of lpragLifLozin treAtment in type2 Diabetes Patients: LONG-TERM (STELLA-LONG TERM)
Brief Title: Specified Drug Use Results Survey of Ipragliflozin Treatment in type2 Diabetes Patients
Acronym: STELLALONGTERM
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SGL002
Record Dates: First submitted 2015-06-15; First posted 2015-06-24 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2018-12

CONDITIONS: Type 2 Diabetes
Keywords: Suglat; SGLT-2 inhibitor; Ipragliflozin L-Proline; ASP1941 long-term use
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suglat group: Tablets
  Interventions: Drug: ipragliflozin

INTERVENTIONS:
Drug: ipragliflozin — Tablets
  Other Names: ASP1941; Suglat

SUMMARY:
The objective of this survey is to confirm the safety of Suglat Tablets

DETAILED DESCRIPTION:
The objective of this survey is to confirm the safety and efficacy of Suglat Tablets for long-term use over 3 years.

Specify the effects of Suglat Tablets on the cardiovascular system, incidence rates of malignant tumor, and their risk factors.

Investigate the occurrence of adverse drug reactions. Specify factors that may possibly influence the safety and efficacy of Suglat Tablets.

<Items of interest>

* Hypoglycemia
* Genital infection
* Urinary tract infection
* Polyuria and pollakiuria
* Adverse events related to a decrease in body fluids (dehydration, etc.)
* Malignant tumor
* Cardiovascular diseases

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes who first use Suglat Tablets during the period from July 17, 2014 to July 16, 2015

Exclusion Criteria:

* off-label use patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes who first use Suglat Tablets during the period from July 17, 2014 to July 16, 2015
Sampling Method: Non-Probability Sample
Enrollment: 11412 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Incidence of cardiovascular adverse events | Up to 3 years
Incidence of malignant tumor | Up to 3 years

SECONDARY OUTCOMES:
Safety developed by adverse events and laboratory tests | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Maegawa H, Tobe K, Nakamura I, Uno S. Real-world evidence for long-term safety and effectiveness of ipragliflozin in treatment-naive versus non-naive Japanese patients with type 2 diabetes mellitus: subgroup analysis of a 3-year post-marketing surveillance study (STELLA-LONG TERM). Diabetol Int. 2021 Mar 24;12(4):430-444. doi: 10.1007/s13340-021-00501-w. eCollection 2021 Oct. PMID 34567926
- [Derived] Nakamura I, Maegawa H, Tobe K, Uno S. Safety and Effectiveness of Ipragliflozin in Elderly Versus Non-elderly Japanese Patients with Type 2 Diabetes: Subgroup Analysis of STELLA-LONG TERM. Diabetes Ther. 2021 May;12(5):1359-1378. doi: 10.1007/s13300-021-01042-w. Epub 2021 Mar 17. PMID 33730336
- [Derived] Maegawa H, Tobe K, Nakamura I, Uno S. Safety and effectiveness of ipragliflozin in elderly versus non-elderly Japanese type 2 diabetes mellitus patients: 12 month interim results of the STELLA-LONG TERM study. Curr Med Res Opin. 2019 Nov;35(11):1901-1910. doi: 10.1080/03007995.2019.1647503. Epub 2019 Aug 29. PMID 31347926
- [Derived] Nakamura I, Maegawa H, Tobe K, Uno S. Safety and Effectiveness of Ipragliflozin for Type 2 Diabetes in Japan: 12-Month Interim Results of the STELLA-LONG TERM Post-Marketing Surveillance Study. Adv Ther. 2019 Apr;36(4):923-949. doi: 10.1007/s12325-019-0895-1. Epub 2019 Feb 14. PMID 30767112
- [Derived] Maegawa H, Tobe K, Tabuchi H, Nakamura I. Baseline characteristics and interim (3-month) efficacy and safety data from STELLA-LONG TERM, a long-term post-marketing surveillance study of ipragliflozin in Japanese patients with type 2 diabetes in real-world clinical practice. Expert Opin Pharmacother. 2016 Oct;17(15):1985-94. doi: 10.1080/14656566.2016.1217994. Epub 2016 Aug 12. PMID 27463414